CLINICAL TRIAL: NCT03339050
Title: Reducing Cardiovascular Risk of Mid-life and Older African Americans
Brief Title: Reducing Cardiovascular Risk of African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Florida A&M University (Other); University of Georgia (Other)
Responsible Party: Principal Investigator, Penny Ralston, Professor and Dean Emeritus, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FloridaStateU
Record Dates: First submitted 2017-07-01; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cardiovascular Risk Factor
Keywords: church-based health promotion; African Americans
MeSH Terms: interventions — Health

STUDY DESIGN:
Intervention Model Description: Health for Hearts United is a longitudinal church-based intervention to reduce cardiovascular disease (CVD) risk in mid-life and older African Americans. Using community-based participatory research (CBPR) approaches and undergirded by both the Transtheoretical Model of Behavior Change and Socio-ecological theory, the 18-month intervention was developed in six North Florida churches (three treatment, three comparison).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health for Hearts United (Experimental): Health for Hearts United (HHU) is a 18-month church-based intervention to reduce CVD risk in mid-life and older African Americans.
  Interventions: Behavioral: Health for Hearts United

INTERVENTIONS:
Behavioral: Health for Hearts United — The intervention was framed around three conceptual components (awareness building, clinical learning, and efficacy development), and four types of programming (church-initiated, joint programming, standard programming (culturally tailored post cards and newsletters), and data collection health promotion (generic materials, clinical sessions with an Registered Dietitian). Key messages were identified for the intervention including eating better, moving around more, reducing stress, and taking charge of your health.

SUMMARY:
Diseases such as hypertension and stroke affect mid-life and older African Americans at higher rates than Whites, negatively affecting health status of this group. This project determine the effectiveness of a faith-based health intervention for mid-life and older African Americans using community-based participatory research approaches.

DETAILED DESCRIPTION:
Mid-life and older African Americans (AAs), a population that is increasing in number, have high rates of cardiovascular-related morbidity and mortality in relation to Whites. For this population, dietary and physical activity behaviors are related to the incidence of cardiovascular disease (CVD). Few tested health promotion interventions tailored for mid-life and older AAs are available yet churches have been shown to be an effective environment for AA health programs. Thus, the overall goal of this project is to reduce CVD risk factors in mid-life and older AAs through implementing and evaluating a church-based health intervention. Using the Transtheoretical Model of Behavior Change (TTM) and Socio-ecological theory (SE), the objectives of this project were to: 1) determine the effectiveness of a church-based intervention in relation to dietary behaviors (food choice, dietary quality), habitual physical activity) and CVD clinical risk factors of mid-life and older African Americans by increasing consumption of fruits, vegetables and calcium-rich foods; decreasing consumption of fat, sugar and sodium; increasing habitual physical activity; and improving selected clinical outcomes (blood pressure, body weight, glucose, among others); 2) identify the differential influence of program components of the intervention; 3) examine variables that might mediate the process of goal achievement; and 4) determine variables that are related to stage of change progression in goal achievement. Midlife and older AAs (n=221) from six churches, three treatment and three comparison, in North Florida were randomly selected from the churches, stratifying by age and gender. The intervention, Health for Hearts United, was developed using a community-based participatory approach and included literature-based conceptual elements of awareness building, clinical learning and efficacy development. Instruments included a food and lifestyle habits questionnaire (food frequency, NCI fruit and vegetable screener, NCI fat screener, physical activity items, TTM items, background characteristics, among others). Clinical data, including 24 hour recall, were collected from a subsample of participants (n=104). Data were collected at four points: Baseline, 6 ,18 and 24 month. The project was guided by research and community advisory committees.

ELIGIBILITY:
Inclusion Criteria:

* 45 years of age or older
* African American
* member and regular attender of church (at least twice a month)
* resident of Gadsden and Leon counties in North Florida.

Exclusion Criteria:

* Under 45 years of age
* not African American
* not a member and regular attender of church
* not a resident of Gadsden and Leon counties in North Florida.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2008-06-03 (Actual); Primary Completion 2013-01-31 (Actual); Study Completion 2013-01-31 (Actual)

PRIMARY OUTCOMES:
Increase in fruit and vegetable consumption assessed by a single item on number of servings of fruits and vegetables consumed daily. | Change from Baseline, 6 months, 18 months and 24 months
  The single item measure was "How many servings of fruits and vegetables do you usually eat each day?" The item had the following possible responses: zero, one, two, three, four, five and six or more servings daily. The range of scores was zero to six, with six representing the highest number of servings daily and zero representing the lowest.
Decrease in saturated fat intake (g) as assessed by the multiple pass 24 hour recall. | Change from Baseline, 6 months, 18 months and 24 months
  The multiple pass 24 hour food recall was taken on three days (two week days and one weekend day) by trained interviewers. Data were analyzed using Food Processor (Esha, Salem, Oregon). The unit of measure was grams (g).
Decrease in total sugar intake (g) as assessed by the multiple pass 24 hour recall. | Change from Baseline, 6 months, 18 months and 24 months
  The multiple pass 24 hour food recall was taken on three days (two week days and one weekend day) by trained interviewers. Data were analyzed using Food Processor (Esha, Salem, Oregon). The unit of measure was grams (g).
Decrease in total sodium intake (g) as assessed by the multiple pass 24 hour recall. | Change from Baseline, 6 months, 18 months and 24 months
  The multiple pass 24 hour food recall was taken on three days (two week days and one weekend day) by trained interviewers. Data were analyzed using Food Processor (Esha, Salem, Oregon). The unit of measure was grams (g).

SECONDARY OUTCOMES:
Increase in habitual physical activity (total kilocalories per week) as assessed by the Yale Physical Activity Scale (YPAS). | Change from Baseline, 6 months, 18 months and 24 months
  The Yale Physical Activity Scale (YPAS) uses a simple checklist to provide estimates of caloric expenditure from activity time (minutes per day or week) and activity dimensions (working, yard work, caretaking, exercising, and recreational activities) during a typical day or week. The unit of measure is kilocalories per week (kcal/week) and is computed by converting all activities into minutes per week, multiplying each by an intensity code for kilocalories, and then summing to determine an energy expenditure summary index (kcal/week). The range of possible scores varies per study but the literature on older adult populations suggests low scores on the YPAS in the 300 kcal/week range and high scores of over 20,000 kcal/week.
Decrease in girth circumference of abdomen (cm) as assessed using clinical measurements by trained staff. | Change from Baseline, 6 months, 18 months and 24 months
  The abdomen was measured in centimeters (cm) with a plastic non-flexible measuring tape (Issaquah, WA). The abdomen was measured at the top of the iliac crest while each participant was exhaling.
Decrease in systolic and diastolic blood pressure (mmHg) as assessed using clinical measurements by trained staff. | Change from Baseline, 6 months, 18 months and 24 months
  Three blood pressure measurements were taken on the non-dominant arm after each participant rested for a few minutes, using a digital device (A&D Medical, Miltitas, CA). The three readings were then averaged. The unit of measure was millimeter of mercury (mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Penny A Ralston, Ph.D., Principal Investigator — Florida State University

IPD SHARING:
Plan to Share IPD: No
We have shared the outcomes of the study through local public events in the local community, invited local presentations, newspaper articles, national refereed presentations, and publications. Publications are already available for researcher use.

REFERENCES:
- [Result] Ralston PA, Lemacks JL, Wickrama KK, Young-Clark I, Coccia C, Ilich JZ, Harris CM, Hart CB, Battle AM, O'Neal CW. Reducing cardiovascular disease risk in mid-life and older African Americans: a church-based longitudinal intervention project at baseline. Contemp Clin Trials. 2014 May;38(1):69-81. doi: 10.1016/j.cct.2014.03.003. Epub 2014 Mar 28. PMID 24685998
- [Result] Ralston PA, Young-Clark I, Coccia C. The Development of Health for Hearts United: A Longitudinal Church-based Intervention to Reduce Cardiovascular Risk in Mid-life and Older African Americans. Ethn Dis. 2017 Jan 19;27(1):21-30. doi: 10.18865/ed.27.1.21. PMID 28115818
- [Result] Wickrama KA, Ralston PA, O'Neal CW, Ilich JZ, Harris CM, Coccia C, Young-Clark I, Lemacks J. Life dissatisfaction and eating behaviors among older African Americans: the protective role of social support. J Nutr Health Aging. 2012;16(9):749-53. doi: 10.1007/s12603-012-0404-6. PMID 23131815
- [Result] O'Neal CW, Wickrama KA, Ralston PA, Ilich JZ, Harris CM, Coccia C, Young-Clark I, Lemacks J. Health insurance status, psychological processes, and older African Americans' use of preventive care. J Health Psychol. 2014 Apr;19(4):491-502. doi: 10.1177/1359105312474911. Epub 2013 Mar 1. PMID 23456216
- [Result] O'Neal CW, Wickrama KK, Ralston PA, Ilich JZ, Harris CM, Coccia C, Young-Clark I, Lemacks J. Eating behaviors of older African Americans: an application of the theory of planned behavior. Gerontologist. 2014 Apr;54(2):211-20. doi: 10.1093/geront/gns155. Epub 2012 Dec 14. PMID 23241919
- [Result] McDole M, Ralston PA, Coccia C, Young-Clark I. The development of a tracking tool to improve health behaviors in African American adults. J Health Care Poor Underserved. 2013 Feb;24(1):171-84. doi: 10.1353/hpu.2013.0003. PMID 23377726
- [Derived] Caffo O, Ralston PA, Lemacks JL, Young-Clark I, Wickrama KKAS, Ilich JZ. Sex and Body Circumferences Associated with Serum Leptin in African American Adults. J Womens Health (Larchmt). 2021 Dec;30(12):1769-1777. doi: 10.1089/jwh.2020.8820. Epub 2021 Mar 3. PMID 33661054
- [Derived] Ralston PA, Wickrama KKAS, Coccia CC, Lemacks JL, Young-Clark IM, Ilich JZ. Health for Hearts United Longitudinal Trial: Improving Dietary Behaviors in Older African Americans. Am J Prev Med. 2020 Mar;58(3):361-369. doi: 10.1016/j.amepre.2019.09.024. Epub 2019 Dec 19. PMID 31866211